CLINICAL TRIAL: NCT06308185
Title: Neonatal Seizures: Correlations Between Clinical and Electroencephalographic Semiology, Etiology, Therapy and Prognosis
Brief Title: Neonatal Seizures: Semiology, Etiology, Therapy and Prognosis Correlations
Status: Active, not recruiting | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: EPINEO
Record Dates: First submitted 2024-03-06; First posted 2024-03-13 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Neonatal Seizure; Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates with seizures: Newborns born at term or prematurely who have had epileptic seizures documented by electroencephalogram in the neonatal period
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — Observational retrospective study on infants with neonatal seizures

SUMMARY:
Epileptic seizures in newborns (often called "neonatal convulsions") represent the most frequent neurological problem in newborns (1-3/1000 newborns). The type of seizure and their etiology is very varied and therefore the therapeutic protocol also requires adaptations with a personalization of the therapeutic approach according to the characteristics of the case according to principles of precision medicine in particular for forms of neonatal epilepsy compared to epileptic seizures acute symptomatic. In recent years it has been highlighted that the clinical characterization and instrumental characterization, in particular electroencephalographic, of epileptic seizures represents an important biomarker that allows the choice of therapy to be oriented appropriately. In the literature there is a lack of single-center studies that relate the type of crisis according to the new ILAE 2017 classification (Fisher 2017) and its proposal for neonatal adaptation (Pressler 2021) with the etiology, type of therapy and outcome neurological after a few years.

The primary aim of the study is to evaluate the correlation between the type of seizure determined according to the ILAE classification (clinical variables), the EEG findings of the epileptic seizures and the specific etiology of the epileptic seizures.

The secondary aim is to evaluate the correlation between seizure type and etiology with effective therapy, length of hospitalization and neurobehavioral development outcome. The study design is a retrospective observational on the population of neonates managed at our center in the last decade.

DETAILED DESCRIPTION:
The clinical and instrumental variables that will be collected are all those relating to the diagnosis and management of neonatal epileptic seizures and the outcome of psychomotor development. The data will be those collected from the electronic medical record. The videoEEG reports will be completed by the re-evaluation of the original EEG tracing, whenever this data is available.

The official ILAE classification of 2017 by Fisher e al. (2017) and the ILAE neonatal adaptation of 2021 by Pressler et al. (2021) will be used for the seizure type classification.

The sample size is estimated at 140 subjects, approximately 10 subjects per year. The extimate derives from the calculation of the average annual incidence of newborns born in our center or transferred from other hospitals in the period 2008-2018.

Since the etiology of neonatal crises is heterogeneous and there are no preliminary scientific data currently available on the topic, it is not possible to calculate exactly a priori the number of subjects necessary for the results to be significant.

The data analysis will be primarily descriptive and epidemiological in order to detect trends in the associations between the variables. Only after this pilot phase will we try, where possible, to apply statistical tests for significance analysis.

At this point, to evaluate the associations between categorical variables (such as between the "seizure type" category and the "etiology" category), where possible, the Chi-square or Fisher test will be used and the odds ratio calculation.

To evaluate the association between quantitative variables such as the association between length of hospital stay and time of instituting the most effective drug from seizure onset (for each specific etiology), linear regression and Pearson correlation will be used. To evaluate the association between categorical variables (predictors) of the neonatal period (such as type of seizure, etiology, etc.) and developmental outcomes expressed as quantitative measures, the Spearman rank correlation test or MANOVA will be used.

ELIGIBILITY:
Inclusion Criteria:

* Neonatal epileptic seizures documented by conventional EEG or amplitude integrated EEG occurring within the interval from 1/1/2009 to 10/31/2022;
* Postmenstrual age at presentation of the seizure: from 23+0 and 44+6 weeks EG;

Exclusion Criteria:

* Patients with a clinical diagnosis of seizures without EEG/aEEG confirmation of seizures.
* Patients who have had epileptic seizures outside the indicated postmenstrual age (from 23+0 up to 44+6)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with epileptic seizures that occurred in the neonatal period, which were confirmed with conventional EEG or aEEG admitted to the Neonatology and Neonatal Intensive Care Unit of Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Seizure Type and etiology correlation | 1 year
  Correlation between seizure type (ILAE classification) and etiology
EEG and etiology correlation | 1 year
  Correlation between EEG background and EEG ictal patterns and etiology

SECONDARY OUTCOMES:
Etiology and and effective drug correlation | 1 year
  Etiology and and effective drug correlation
Etiology and neurobehavioral outcome correlation | 1 year
  Correlation etiology and neurobehavioral outcome determined the neurological examination and neurodevelopmental test at follow up

CONTACTS AND LOCATIONS:
Overall Officials: Robertino Dilena, MD, Principal Investigator — Fondazione IRCCS C' Granda Ospedale Maggiore Policlinico
Locations (1):
- Fondazione IRCSS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pisani F, Facini C, Bianchi E, Giussani G, Piccolo B, Beghi E. Incidence of neonatal seizures, perinatal risk factors for epilepsy and mortality after neonatal seizures in the province of Parma, Italy. Epilepsia. 2018 Sep;59(9):1764-1773. doi: 10.1111/epi.14537. Epub 2018 Aug 22. PMID 30132843
- [Result] Cornet MC, Sands TT, Cilio MR. Neonatal epilepsies: Clinical management. Semin Fetal Neonatal Med. 2018 Jun;23(3):204-212. doi: 10.1016/j.siny.2018.01.004. Epub 2018 Jan 31. PMID 29426806
- [Result] Nunes ML, Yozawitz EG, Zuberi S, Mizrahi EM, Cilio MR, Moshe SL, Plouin P, Vanhatalo S, Pressler RM; Task Force on Neonatal Seizures, ILAE Commission on Classification & Terminology. Neonatal seizures: Is there a relationship between ictal electroclinical features and etiology? A critical appraisal based on a systematic literature review. Epilepsia Open. 2019 Jan 25;4(1):10-29. doi: 10.1002/epi4.12298. eCollection 2019 Mar. PMID 30868112
- [Result] Shellhaas RA, Wusthoff CJ, Tsuchida TN, Glass HC, Chu CJ, Massey SL, Soul JS, Wiwattanadittakun N, Abend NS, Cilio MR; Neonatal Seizure Registry. Profile of neonatal epilepsies: Characteristics of a prospective US cohort. Neurology. 2017 Aug 29;89(9):893-899. doi: 10.1212/WNL.0000000000004284. Epub 2017 Jul 21. PMID 28733343
- [Result] Fisher RS, Cross JH, French JA, Higurashi N, Hirsch E, Jansen FE, Lagae L, Moshe SL, Peltola J, Roulet Perez E, Scheffer IE, Zuberi SM. Operational classification of seizure types by the International League Against Epilepsy: Position Paper of the ILAE Commission for Classification and Terminology. Epilepsia. 2017 Apr;58(4):522-530. doi: 10.1111/epi.13670. Epub 2017 Mar 8. PMID 28276060
- [Result] Pressler RM, Cilio MR, Mizrahi EM, Moshe SL, Nunes ML, Plouin P, Vanhatalo S, Yozawitz E, de Vries LS, Puthenveettil Vinayan K, Triki CC, Wilmshurst JM, Yamamoto H, Zuberi SM. The ILAE classification of seizures and the epilepsies: Modification for seizures in the neonate. Position paper by the ILAE Task Force on Neonatal Seizures. Epilepsia. 2021 Mar;62(3):615-628. doi: 10.1111/epi.16815. Epub 2021 Feb 1. PMID 33522601